CLINICAL TRIAL: NCT00370370
Title: Intravitreal Bevacizumab vs. Bevacizumab Combined With Triamcinolone for Neovascular AMD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8533
Record Dates: First submitted 2006-08-30; First posted 2006-08-31 (Estimated); Last update posted 2008-06-26 (Estimated); Status verified 2008-06

CONDITIONS: Neovascular Age-Related Macular Degeneration
Keywords: Bevacizumab,; Triamcinolone; Age-related macular degeneration; Choroidal neovascular membrane
MeSH Terms: conditions — Macular Degeneration | interventions — Bevacizumab; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Active Comparator): Injection of intravitreal bevacizumab
  Interventions: Drug: bevacizumab
- 2 (Active Comparator): Injection of bevacizumab + triamcinolone acetonide
  Interventions: Drug: bevacizumab + triamcinolone acetonide

INTERVENTIONS:
Drug: bevacizumab — Injection of intravitreal bevacizumab
  Arms: 1
Drug: bevacizumab + triamcinolone acetonide — Injection of bevacizumab + triamcinolone acetonide
  Arms: 2

SUMMARY:
To compare the efficacy and safety results of intravitreal bevacizumab alone with bevacizumab + triamcinolone acetonide in neovascular AMD.

ELIGIBILITY:
Inclusion Criteria:

* Cases of active neovascular AMD with visual acuity of 20/400- 20/40

Exclusion Criteria:

* History of glaucoma or ocular hypertension
* Disciform scar

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-11

PRIMARY OUTCOMES:
visual acuity

SECONDARY OUTCOMES:
central macular thickness
leakage in fluorescein angiography
intraocular pressure
anterior chamber reaction

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Ahmadieh, MD, Principal Investigator — Ophthalmic Research Center of Shaheed Beheshti Medical University
Locations (1):
- Hamid Ahmadieh, MD, Tehran, Tehran Province, Iran